CLINICAL TRIAL: NCT06156774
Title: SARcopenia and Simplified Geriatric Assessment in Lymphoma Patients Undergoing CAR-T Cell Therapy: the FIL_SAR-CAR Project
Status: Recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Other Study IDs: FIL_SAR-CAR
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Non-hodgkin Lymphoma,B Cell
Keywords: Non-hodgkin Lymphoma,B Cell; CAR-T; Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Immunotherapy, Adoptive; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Non-Hodgkin Lymphoma B cell: Patients with B-cell non-Hodgkin Lymphoma scheduled to received CAR-T cell product according to Agenzia Italiana del Farmaco (AIFA) indications and technical data sheet of the drug
  Interventions: Other: Chimeric Antigen Receptor T-cells (CAR-T) therapy

INTERVENTIONS:
Other: Chimeric Antigen Receptor T-cells (CAR-T) therapy — Patients will be treated with CAR-T cell product as per routine clinical practice.

SUMMARY:
This is a multicenter prospective observational study lead by the FIL on sarcopenia and sGA as possible predictors of efficacy and toxicity outcomes in patients undergoing CAR-T cells treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old).
* Patients with B-cell non-Hodgkin Lymphoma scheduled to received CAR-T cell product according to Agenzia Italiana del Farmaco (AIFA) indications and technical data sheet of the drug
* Availability of a 18F-FDG PET/CT scan or a full dose CT scan (without contrast media) pre-treatment with CART
* Written informed consent voluntarily provided

Exclusion Criteria:

* Patients not fulfilling the eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with B-cell non-Hodgkin Lymphoma scheduled to received CAR-T cell product according to Agenzia Italiana del Farmaco (AIFA) indications and technical data sheet of the drug
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response Rates (ORR) | up to 28 months
  Best Overall Response Rates (ORR) after CAR-T therapy according to the presence or absence of sarcopenic status

SECONDARY OUTCOMES:
Best Complete Remission Rates (CRR) | up to 28 months
  Best Complete Remission Rates (CRR) after CAR-T therapy
Progression-Free Survival (PFS) | up to 28 months
  Progression-Free Survival (PFS) at + 12 months after CAR-T therapy
Overall Survival (OS) | up to 28 months
  Overall Survival (OS) at + 12 months after CAR-T therapy
Incidence of CAR-T related toxicities | up to 28 months
  Incidence of CAR-T related toxicities (specifically: CRS, ICANS, cytopenias) in the different sarcopenic subgroups and, for patients ≥65 years old, according to their functional status
Rate of admission to Intensive Care Units (ICU) | up to 28 months
  Rate of admission to Intensive Care Units (ICU) according to patients' sarcopenic and functional status

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Ruggero Zilioli, Principal Investigator — ASST Grande Ospedale Metropolitano Niguarda, Milano, Italy
Locations (21):
- Italy (21):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo - S.C.D.U. Ematologia, Alessandria
  - AOU Ospedali Riuniti - Clinica di Ematologia, Ancona
  - Azienda Ospedaliera S .Giuseppe Moscati - S.C. Ematologia e Trapianto emopoietico, Avellino
  - IRCCS Centro di Riferimento Oncologico di Aviano - Divisione di Oncologia e dei Tumori immuto-correlati, Aviano
  - ASST Spedali Civili di Brescia - S.C. Ematologia, Brescia
  - Ospedale di Castelfranco Veneto - Oncoematologia IOV, Castelfranco Veneto
  - Azienda Ospedaliera Universitaria Careggi - Unità funzionale di Ematologia, Florence
  - ASST Grande Ospedale Metropolitano Niguarda - S.C. Ematologia, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano - Ematologia, Milan
  - Istituto Scientifico San Raffaele - Unità Linfomi - Dipartimento Oncoematologia, Milan
  - A.O. Ospedali Riuniti Villa Sofia-Cervello - Divisione di Ematologia, Palermo
  - Ospedale S. Maria della Misericordia - Ematologia, Perugia
  - Ospedale Guglielmo da Saliceto - U.O. Ematologia, Piacenza
  - AOU Pisana - U.O. Ematologia, Pisa
  - Azienda Unità Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia, Reggio Emilia
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Università Cattolica S. Cuore - Ematologia, Roma
  - Policlinico Umberto I - Università "La Sapienza" - Istituto Ematologia -Dipartimento di Medicina Traslazionale e di Precisione, Roma
  - A.O.U. Citta della Salute e della Scienza di Torino - S.C. Ematologia, Torino
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC) - Clinica di Ematologia, Udine
  - AOU Integrata di Verona - U.O. Ematologia, Verona
  - ULSS 8 Berica - Ospedale S. Bortolo - Ematologia, Vicenza